CLINICAL TRIAL: NCT06130228
Title: Multi-ingredient Supplementation as an Adjunctive Therapy in Late-onset Pompe Disease
Brief Title: Nutritional Therapy in Late-onset Pompe Disease
Acronym: PDT-MIS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Mark Tarnopolsky, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17004
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Pompe Disease; Muscle Loss; Obesity; Nutrition Poor; Lysosomal Storage Diseases; Glycogen Storage Disease Type II; Glycogen Storage Disease Type II Late Onset; Glycogen Storage Disease Type II, Adult
Keywords: Muscle; Supplements; Antioxidants; Whey; Casein; Vitamin D; Creatine; Calcium; Omega-3; Green coffee bean; Green tea; CoQ10; Alpha-lipoic acid; Vitamin E; Weight loss; Obesity; Muscle strength; 6-meter walk test; Pompe disease; Oxidative stress; Mitochondria; Autophagy; Glycogen; Forskolin; Beet root; Performance
MeSH Terms: conditions — Glycogen Storage Disease Type II; Muscular Atrophy; Obesity; Malnutrition; Lysosomal Storage Diseases; Weight Loss

STUDY DESIGN:
Intervention Model Description: The present study is a 4-month randomized double-blind, placebo controlled, clinical trial with two treatments arms and groups (PDT-MIS and PLA).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Following medical screening and consent, all patients accepted into the study will be assigned a unique identifier number (1-28), which will be provided to an outside party not associated with Dr. Tarnopolsky or co-investigators that will randomize each subject to one of two experimental conditions. Dr. Tarnopolsky, co-investigators, and the subjects will be blinded to the treatment allocations for the duration of the 4-month trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-ingredient supplement (PDT-MIS) (Experimental): Multi-ingredient supplementation (PDT-MIS) consists of daily intake of high-quality proteins, creatine, vitamin D, calcium, plant extracts (green coffee bean, green tea, beet root, and forskolin), and Omega-3 fatty acids. Concurrent with supplementation, patients will do mixed rehabilitative exercise (cardio and strength) and respiratory muscle training four days a week.
  Interventions: Dietary Supplement: Multi-ingredient supplement (PDT-MIS)
- Placebo (PLA) (Placebo Comparator): Placebo (PLA) consists of daily intake of collagen, safflower, and microcrystalline cellulose. Concurrent with supplementation, patients will do mixed rehabilitative exercise (cardio and strength) and respiratory muscle training four days a week.
  Interventions: Dietary Supplement: Placebo (PLA)

INTERVENTIONS:
Dietary Supplement: Multi-ingredient supplement (PDT-MIS) — Supplementation with active PDT-MIS daily
  Arms: Multi-ingredient supplement (PDT-MIS)
Dietary Supplement: Placebo (PLA) — Supplementation with inactive placebo
  Arms: Placebo (PLA)

SUMMARY:
RATIONALE: Pompe disease (PD) is a recessive genetic disorder wherein the body cannot break down glycogen due to a mutation in the acid alpha glucosidase (GAA) gene, which encodes for acid alpha-glucosidase. The adult/late onset form (LOPD) leads to glycogen accumulation and autophagic buildup, causing progressive muscle weakness that leads to wheelchair dependence, reduced quality of life and premature death due to cardiorespiratory insufficiency. While nutritional strategies, such as the low carbohydrate/high protein and ketogenic diets, have been used clinically, they are difficult to maintain and have limited benefits. Multi-ingredient supplementation (MIS) allows for targeting of several underlying pathogenic pathways and may be more convenient than traditional dietary strategies, thereby improving both adherence and LOPD pathology.

DETAILED DESCRIPTION:
DESIGN AND INTERVENTION: The present study is a 4-month randomized, double-blind, placebo-controlled clinical trial (RCT) with sampling pre and post intervention in late onset Pompe disease patients undergoing enzyme replacement therapy (ERT) (21-90 years of age). Each patient will be randomized into either a Pompe-Targeted Multi-Ingredient Supplement (PDT-MIS; high-quality proteins, antioxidants, plant extracts, vitamins, and omega-3 fatty acids,) or placebo (PLA; collagen, safflower, and cellulose) group and then undergo four months of daily supplementation with concurrent rehabilitative exercise training (mixed cardio and strength four days/week) and respiratory muscle training (four days/week).

GENERAL RESEARCH AIMS AND HYPOTHESIS: The purpose of this study is to investigate the benefits of PDT-MIS on muscle and blood pathology, muscle function, respiratory capacity, and health-related quality of life (HRQOL) in LOPD patients on enzyme replacement therapy (ERT). It is generally hypothesized that PTD-MIS will mitigate mitochondrial dysfunction, oxidative damage, inflammation and alleviate 'autophagic block' in skeletal muscle of LOPD patients. PDT-MIS may therefore improve muscle pathology by affecting several cell pathways simultaneously, and thereby enhance muscle function, respiratory capacity, and HRQOL of LOPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed LOPD
* Have undergone enzyme replacement therapy for at least three months.
* Physically capable of doing rehabilitative exercise, respiratory muscle training, and the clinical tests described herein.

Exclusion Criteria:

* Dairy protein allergy
* Renal disease (creatinine > 140)
* Attempting pregnancy or currently pregnant
* Current supplementation

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in the body composition index by DEXA analyses | Baseline to 4 months
  Body composition index (lean mass/fat mass ratio)
Percent change in seated pulmonary function by spirometry | Baseline to 4 months
  Seated forced expiratory volume/forced vital capacity ratio (FEV1/FVC)
Percent change in supine pulmonary function by spirometry | Baseline to 4 months
  Supine forced expiratory volume/forced vital capacity ratio (FEV1/FVC)
Percent change in 6-minute walking test distance | Baseline to 4 months
  6-minute walking test distance (meters)

SECONDARY OUTCOMES:
Percent change in health-related quality of life by SF-36 Survey | Baseline to 4 months
  36-item short form survey (ranging from low 0 to high 100)
Percent change in health-related quality of life by Rotterdam Handicap Score | Baseline to 4 months
  Rotterdam Handicap Score (ranging from low 9 to high 36)
Percent change in health-related quality of life by the R-Pact Questionnaire | Baseline to 4 months
  Rasch-built Pompe-specific Activity (ranging from low 0 to high 100 points)
Percent change in maximal grip strength by dynamometry | Baseline to 4 months
  Maximal grip strength (kilogram)
Percent change in isometric leg strength by Biodex | Baseline to 4 months
  Isometric leg strength (newton meters)
Percent change in leg strength by 4-step stair climb test | Baseline to 4 months
  4-step stair climb time (seconds)
Percent change in lower extremity functioning by short physical performance battery (SPPB) | Baseline to 4 months
  Short physical performance battery (ranging from low 0 to high 12)
Percent change in lower extremity functioning by timed get up and go test (TUG) | Baseline to 4 months
  Timed get up and go test (seconds)
Percent change in total muscle glycogen by ELISA | Baseline to 4 months
  Total muscle glycogen (ug per mg of tissue)
Percent change in lysosomal glycogen in muscle by high-resolution light microscopy | Baseline to 4 months
  Lysosomal glycogen (% total muscle area)
Percent change in autophagic area in muscle by electron microscopy | Baseline to 4 months
  Autopgahic area (% total muscle area)
Percent change in p62 expression in muscle by Western blotting | Baseline to 4 months
  p62 expression (optical density)
Percent change in complex I-V expression in muscle by Western blotting | Baseline to 4 months
  Complex I-V expression (optical density)
Percent change in 4-hydroxynonenal levels in muscle by Western blotting | Baseline to 4 months
  4-hydroxynonenal levels (optical density)
Percent change in galactin-3 expression in muscle by Western blotting | Baseline to 4 months
  Galactin-3 expression (optical density)
Percent change in superoxide dismutase 1 expression in muscle by Western blotting | Baseline to 4 months
  Superoxide dismutase 1 expression (optical density)
Percent change in superoxide dismutase 2 expression in muscle by Western blotting | Baseline to 4 months
  Superoxide dismutase 2 expression (optical density)

OTHER OUTCOMES:
Percent change in malondialdehyde levels in blood | Baseline to 4 months
  Malondialdehyde levels (ng/mL)
Percent change in Oxygen Radical Absorbance Capacity in blood | Baseline to 4 months
  Oxygen Radical Absorbance Capacity (relative fluorescence units)
Percent change in interleukin 6 levels in blood | Baseline to 4 months
  interleukin 6 levels (pg/dL)
Percent change in interleukin 1 levels in blood | Baseline to 4 months
  interleukin 1 levels (pg/dL)
Percent change in interleukin 10 levels in blood | Baseline to 4 months
  interleukin 10 levels (pg/dL)
Percent change in tumor necrosis factor alpha levels in blood | Baseline to 4 months
  tumor necrosis factor alpha (pg/dL)
Percent change in c-reactive protein levels in blood | Baseline to 4 months
  c-reactive protein levels (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Tarnopololsky, MD/PhD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No